CLINICAL TRIAL: NCT03797534
Title: Individualized Administration of Warfarin by Polymorphisms of VKORC1 and CYP2C9 Genes:A Randomized Controlled Trial, Multi-center Trial
Brief Title: Individualized Administration of Warfarin by Polymorphisms of VKORC1 and CYP2C9 Genes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Liang-Wan Chen MD, The director of the department of cardiovascular surgery, Fujian Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CLW2018WA
Record Dates: First submitted 2019-01-06; First posted 2019-01-09 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Heart Valve Prosthesis
Keywords: warfarin; gene

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard anticoagulant group (No Intervention)
- Bayesian model group (Experimental)
  Interventions: Other: dose regime

INTERVENTIONS:
Other: dose regime — The initial dose of the experimental group will be calculated by the Bayesian model.
  Arms: Bayesian model group

SUMMARY:
The purpose of this study is to explore the individualized administration model of warfarin suitable for Chinese people, and provide a scientific reference for the use of warfarin to Chinese people.

DETAILED DESCRIPTION:
About 600 patients with VKORC1 and CYP2C9 gene mutations were included in the treatment of warfarin anticoagulant therapy. The main indications include valve replacement, atrial fibrillation, pulmonary embolism, etc., randomly divided into 2 groups, respectively, the control group (that is, the use of fixed-dose group), Bayesian-model group, the use of single-blind treatment method, to evaluate the number of major adverse events, TTR and INR adjustments in patients between different groups after three months of taking warfarin, and then to explore the individualized drug use model of warfarin suitable for Chinese population.

In the Bayesian group, according to the genotype of VKORC1 and CYP2C9, the stable dose was calculated by the dose prediction model of Bayesian, and the first three drugs were taken at this dose, and then adjusted to the actual stable dose according to the change of INR. Meanwhile, the control group was administered according to the traditional way, that is, the initial dose is 2.5 or 3mg/d and is gradually adjusted to a stable dose according to changes of INR. The monitoring frequency of INR is: once a day from the beginning of the drug to the time of discharge, once a week after discharge, and once a month after the stable dose is obtained. Detailed records of the number of days to reach a stable dose, the INR value and the occurrence of side effects and time are documented. The concrete steps are as follows:

1. clinicians to judge the standard of the selection criteria;
2. to obtain the consent of the patient and sign an informed consent certificate;
3. to collect 2ml anticoagulant blood before the drug, fill in the application form for individualized drug use in warfarin, and indicate the experimental group and control group;
4. the specimen assigned to the laboratory for Genotyping;
5. lab to calculate the predicted stable warfarin dose and the results fed back to the clinician within one working day after receiving the specimen;
6. in the control group, the drug retained at the regular dose, and the first 3 days of the experimental group administered at the predicted dose;
7. the dosage of warfarin in the two groups of cases adjusted to the stable dose according to the value, and the adjustment amplitude of the experimental group also referred to the predicted stable dose.
8. to monitor INR once a day during hospitalization, and to those who do not receive a stable dose of discharge, follow up and monitor INR once a week until a stable dose or medication is obtained for 90 days;
9. to document clinical trial records, including the daily use of warfarin, each detection of the appearance of the situation like INR value, bleeding, venous embolism and other side effects.

Finally，according to the outcome parameters,statistical analysis were performed with SPSS 11.5 software. A value of P < 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 14 years old；
2. Warfarin anticoagulant therapy is required for at least 3 months；
3. The genotype of patient VKORC1 is non-AA, CYP2C9 genotype is non*1/*1； the patients who are followed up, regularly monitored for INR and willing to provide peripheral blood for DNA extraction and genetic testing；
4. The patient or family members can understand the research plan and will participate in this study and provide a written informed consent；

Exclusion Criteria:

1. Severe liver dysfunction (ChildPugh ≥ 10);
2. Severe infection, respiratory failure;
3. Severe heart failure ( NYHA ≥ IV);
4. Severe renal insufficiency (Ccr ≤ 20ml / min);
5. Cancer;
6. Diseases of the blood system;
7. Severe pulmonary hypertension (PAPm ≥ 45mmHg);
8. Abnormal thyroid function;
9. Patients with a history of venous thromboembolism, or serious events such as severe bleeding or embolism;
10. Women who are pregnant or breastfeeding;
11. Taking or planning to take other oral anticoagulants;
12. The base INR value is >1.4;
13. VKORC1, CYP2C9 genotypes are AA, *1/*1;
14. Secondary valve replacement surgery;
15. Emergency hospital admission for valve surgery;
16. Diagnosis of coronary atherosclerotic heart disease;
17. Severe mental illness, mental disorder ; -

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2019-02-01 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
excessive anticoagulant time ratio | 3 months postoperatively
  INR>3，INR>4
The occurrence of primary bleeding events | 3 months postoperatively
  gastrointestinal hemorrhage, intracerebral hemorrhage,etc
The occurance of secondary bleeding events | 3 months postoperatively
  nasal bleeding, skin stasis,etc
The occurrence of thrombosis events | 3 months postoperatively
  ischemic stroke, deep vein thrombosis,etc

SECONDARY OUTCOMES:
Percentage of time in therapeutic range | 3 months, 6 months, 12 months postoperatively
The time required to reach the treatment target INR for the first time; | 3 months postoperatively
The time required from the beginning of treatment to the stable dose; | 3 months postoperatively
The percentage of time below the target INR range; | 3 months postoperatively
The percentage of time above the target INR range; | 3 months postoperatively
The number of dose adjustments and the number of INR measured during the first month of treatment; | 3 months postoperatively
The proportion of patients in each group receiving a stable dose after follow-up; | 3 months postoperatively
The proportion of patients in each group having side effects after follow-up | 3 months postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- the Department of Cardiovascular Surgery, Fuzhou, Fujian, China

REFERENCES:
- [Background] Gage BF, Eby C, Johnson JA, Deych E, Rieder MJ, Ridker PM, Milligan PE, Grice G, Lenzini P, Rettie AE, Aquilante CL, Grosso L, Marsh S, Langaee T, Farnett LE, Voora D, Veenstra DL, Glynn RJ, Barrett A, McLeod HL. Use of pharmacogenetic and clinical factors to predict the therapeutic dose of warfarin. Clin Pharmacol Ther. 2008 Sep;84(3):326-31. doi: 10.1038/clpt.2008.10. Epub 2008 Feb 27. PMID 18305455
- [Background] International Warfarin Pharmacogenetics Consortium; Klein TE, Altman RB, Eriksson N, Gage BF, Kimmel SE, Lee MT, Limdi NA, Page D, Roden DM, Wagner MJ, Caldwell MD, Johnson JA. Estimation of the warfarin dose with clinical and pharmacogenetic data. N Engl J Med. 2009 Feb 19;360(8):753-64. doi: 10.1056/NEJMoa0809329. PMID 19228618
- [Background] Hamberg AK, Hellman J, Dahlberg J, Jonsson EN, Wadelius M. A Bayesian decision support tool for efficient dose individualization of warfarin in adults and children. BMC Med Inform Decis Mak. 2015 Feb 7;15:7. doi: 10.1186/s12911-014-0128-0. PMID 25889768
- [Background] Pirmohamed M, Burnside G, Eriksson N, Jorgensen AL, Toh CH, Nicholson T, Kesteven P, Christersson C, Wahlstrom B, Stafberg C, Zhang JE, Leathart JB, Kohnke H, Maitland-van der Zee AH, Williamson PR, Daly AK, Avery P, Kamali F, Wadelius M; EU-PACT Group. A randomized trial of genotype-guided dosing of warfarin. N Engl J Med. 2013 Dec 12;369(24):2294-303. doi: 10.1056/NEJMoa1311386. Epub 2013 Nov 19. PMID 24251363
- [Background] Kimmel SE, French B, Kasner SE, Johnson JA, Anderson JL, Gage BF, Rosenberg YD, Eby CS, Madigan RA, McBane RB, Abdel-Rahman SZ, Stevens SM, Yale S, Mohler ER 3rd, Fang MC, Shah V, Horenstein RB, Limdi NA, Muldowney JA 3rd, Gujral J, Delafontaine P, Desnick RJ, Ortel TL, Billett HH, Pendleton RC, Geller NL, Halperin JL, Goldhaber SZ, Caldwell MD, Califf RM, Ellenberg JH; COAG Investigators. A pharmacogenetic versus a clinical algorithm for warfarin dosing. N Engl J Med. 2013 Dec 12;369(24):2283-93. doi: 10.1056/NEJMoa1310669. Epub 2013 Nov 19. PMID 24251361
- [Background] Li X, Yang J, Wang X, Xu Q, Zhang Y, Yin T. Clinical benefits of pharmacogenetic algorithm-based warfarin dosing: meta-analysis of randomized controlled trials. Thromb Res. 2015 Apr;135(4):621-9. doi: 10.1016/j.thromres.2015.01.018. Epub 2015 Jan 17. PMID 25628141